CLINICAL TRIAL: NCT04456998
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Clinical Study to Evaluate the Efficacy and Safety of Oral Inhalation of GB002 for the Treatment of WHO Group 1 Pulmonary Arterial Hypertension (PAH)
Brief Title: GB002 in Adult Subjects With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GB002, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB002-2101
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Artery Hypertension
Keywords: seralutinib
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects, investigators, other site personnel, and Sponsor (and/or designee) personnel who are directly involved in the conduct of the study, collection of the data, and analysis of the final safety and efficacy results will remain blinded to treatment assignments until after the completion of the study and the database has been locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- GB002 (seralutinib) (Experimental): GB002 (seralutinib) inhaled orally twice per day (BID) for 24 weeks
  Interventions: Drug: GB002 (seralutinib); Device: Generic Dry Powder Inhaler
- Placebo (Placebo Comparator): Placebo inhaled orally BID for 24 weeks
  Interventions: Drug: Placebo; Device: Generic Dry Powder Inhaler

INTERVENTIONS:
Drug: GB002 (seralutinib) — Capsule containing GB002 (seralutinib)
  Arms: GB002 (seralutinib)
Drug: Placebo — Matching capsule containing placebo
  Arms: Placebo
Device: Generic Dry Powder Inhaler — Generic dry powder inhaler for GB002 (seralutinib) or placebo delivery

SUMMARY:
The primary objective for this trial is to determine the effect of GB002 (seralutinib) on improving pulmonary hemodynamics in subjects with World Health Organization (WHO) Group 1 PAH who are Functional Class (FC) II and III. The secondary objective for this trial is to determine the effect of GB002 (seralutinib) on improving exercise capacity in this population.

ELIGIBILITY:
Inclusion Criteria:

1. A current diagnosis of symptomatic PAH classified by one of the following:

   1. Idiopathic PAH (IPAH) or heritable pulmonary arterial hypertension (HPAH).
   2. PAH associated with connective tissue disease (CTD-APAH).
   3. PAH associated with anorexigen or methamphetamine use.
   4. Congenital heart disease with simple systemic to pulmonary shunt at least 1 year after surgical repair.
2. 6MWD ≥ 150 meters and ≤ 550 meters at screening.
3. WHO FC II or III symptomatology.
4. Treatment with standard of care PAH background therapies.
5. Documentation of cardiac catheterization within the screening period that is consistent with the diagnosis of PAH and meeting all the following criteria, to be confirmed by a central hemodynamic core laboratory:

   1. Mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg (at rest), AND
   2. PVR ≥ 400 dyne•sec/cm5, AND
   3. Pulmonary capillary wedge pressure (PCWP) or left ventricular-end diastolic pressure (LVEDP) ≤12 mm Hg if PVR ≥400 to <500 dyne∙sec/cm5 OR
   4. PCWP or LVEDP ≤15 mmHg if PVR ≥500 dyne∙sec/cm5
6. Pulmonary function tests (PFTs) at screening with the following criteria met:

   1. Forced expiratory volume in 1 second (FEV1) divided by the forced vital capacity (FVC) ≥70%;
   2. Total lung capacity (TLC) or FVC ≥ 70% predicted

Exclusion Criteria:

1. Evidence of chronic thromboembolic disease or acute pulmonary embolism as assessed by ventilation-perfusion (V/Q) scan, computed tomography (CT)-angiogram, or pulmonary angiogram prior to screening.
2. Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure > 160 mm Hg or sitting diastolic blood pressure > 100 mm Hg during screening visit after a period of rest.
3. Systolic blood pressure < 90 mm Hg during screening and baseline visits.
4. WHO Pulmonary Hypertension Group 2-5.
5. Human immunodeficiency virus (HIV)-associated PAH.
6. History of left-sided heart disease and/or clinically significant cardiac disease.
7. Untreated severe obstructive sleep apnea.
8. History of atrial septostomy within 180 days prior to screening.
9. Pulmonary venous occlusive disease (PVOD).
10. Subjects with a history of portopulmonary hypertension or portal hypertension due to cirrhosis classified as Child-Pugh Class A or higher; or baseline ALT or AST > 2 x ULN or Total Bilirubin ≥ 2 x ULN.
11. History of malignancy within 5 years prior to screening.
12. History of a potentially life-threatening cardiac arrhythmia with an ongoing risk.
13. Severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or IP administration (eg; history intracranial hemorrhage).
14. Chronic renal insufficiency as defined by an estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2 via Chronic Kidney Disease Epidemiology Collaboration (CKD-epi) at screening or requires dialytic therapy or hemofiltration.
15. Hemoglobin (Hgb) concentration < 8.5 g/dL at screening.
16. Evidence of active HIV, Hepatitis B or Hepatitis C, or tuberculosis (TB) infections.
17. Inhaled prostanoids; these drugs may be withdrawn ≥ 4 weeks prior to or at screening, if clinically indicated.
18. Use of oral anticoagulants (ie, warfarin or NOAC) at randomization.
19. Requirement of intravenous (IV) inotropes (ie, levosimendan, dopamine, dobutamine, milrinone, norepinephrine) other than an IV prostanoid within 4 weeks of screening.
20. Prior participation in GB002 studies and/or prior treatment with GB002.
21. Currently participating in or has participated in a study of an investigational agent or has used an investigational device for the treatment of PAH within 4 weeks prior to screening.
22. Current use of inhaled tobacco and/or inhaled marijuana.
23. Current alcohol use disorder as defined by DSM-5 and/or positive test for drugs of abuse (amphetamines, methamphetamines, cocaine, phencyclidine [PCP]).
24. Subjects with a history of severe milk protein allergy. In addition, subjects with known intolerance or hypersensitivity to lactose who, in the opinion of the investigator, may experience severe symptoms following the ingestion of lactose.
25. QTcF of > 480 msec recorded on a screening or baseline ECG or receiving concurrent treatment with medications that prolong QT interval.
26. Have any other condition or reason that, in the opinion of the Investigator or Medical Monitor, would prohibit the subject from participating in the study.

NOTE: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aranda, Study Director — Gossamer Bio Inc.
Locations (63):
- United States (36):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Dept of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - The University of California San Francisco, San Francisco, California
  - Medical Corporation, Santa Barbara, California
  - Stanford Healthcare, Stanford, California
  - The Lundquist Institute of Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Central Florida Pulmonary Group, PA, Altamonte Springs, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The Emory Clinic, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Research Center, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (4):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St Vincent's Hospital Melbourne, Fitzroy
  - Royal Hobart Hospital, Hobart
  - Westmead Hospital, Westmead
- Austria (2):
  - LKH - Univ. Klinikum Graz - Universitatsklinik fur Innere Medizin, Graz
  - Medizinische Universitat Wien - Universitatsklinik fur Innere Medizin II, Vienna
- Belgium (2):
  - Erasme University Hospital, Brussels
  - University Hospital of Leuven, Leuven
- Canada (3):
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - Peter Lougheed Centre, Calgary
  - London Health Sciences Centre - Victoria Hospital, London
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- France (2):
  - AP-HP, Hopital de Bicetre, Le Kremlin-Bicêtre
  - CHU de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
- Germany (6):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - DRK Kliniken Berlin - Westend, Berlin
  - Universitätsklinikum Giessen / Marburg, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Zentrum fur Pulmonale Hypertonie Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Universitatsklinikum Regensburg, Regensburg
- Serbia (2):
  - University Clinical Centre of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation, Cambridge
  - Imperial College Healthcare NHS Trust - Hammersmith Medicines Research Limited, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frantz RP, McLaughlin VV, Sahay S, Escribano Subias P, Zolty RL, Benza RL, Channick RN, Chin KM, Hemnes AR, Howard LS, Sitbon O, Vachiery JL, Zamanian RT, Cravets M, Roscigno RF, Mottola D, Osterhout R, Bruey JM, Elman E, Tompkins CA, Parsley E, Aranda R, Zisman LS, Ghofrani HA; TORREY Study Investigators. Seralutinib in adults with pulmonary arterial hypertension (TORREY): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Respir Med. 2024 Jul;12(7):523-534. doi: 10.1016/S2213-2600(24)00072-9. Epub 2024 May 2. PMID 38705167

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo inhaled orally twice per day (BID) for 24 weeks
- GB002 (Seralutinib): GB002 (seralutinib) inhaled orally BID for 24 weeks
Period: Overall Study
Arm/Group | Placebo | GB002 (Seralutinib)
Started | 42 | 44
Completed | 42 | 38
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Protocol Deviation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GB002 (Seralutinib) | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.81) | 48.3 (12.70) | 48.8 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 37 | 37 | 74
  Black or African American | 1 | 0 | 1
  Asian | 2 | 4 | 6
  Other, Not Specified | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 34 | 36 | 70
  Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Pulmonary Vascular Resistance (PVR)
Description: PVR was evaluated using right heart catheterization (RHC).
Time Frame: Baseline, Week 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: dyne•s/cm^5
Arm/Group | Placebo | GB002 (Seralutinib)
Number analyzed (Participants) | 42 | 44
dyne•s/cm^5 | 21.2 [-37.4 to 79.8] | -74.9 [-139.7 to -10.2]
Statistical Analysis 1: Comparison: Placebo vs GB002 (Seralutinib); Test type: Superiority; p = 0.0310, ANCOVA; Mean Difference (Net) = -96.1, 95% CI 2-sided [-183.5 to -8.8] — GB002 vs. Placebo

2. Secondary Outcome: Change From Baseline to Week 24 in Distance Achieved on the Six-Minute Walk Test (6MWT)
Description: The 6MWT measures the distance a participant is able to walk quickly on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline, Week 24
Population: ITT Population: all participants who were randomized. Participants with a baseline and post-baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Placebo | GB002 (Seralutinib)
Number analyzed (Participants) | 42 | 38
meters | 7.4 [-11.2 to 25.9] | 13.9 [-5.1 to 32.8]
Statistical Analysis 1: Comparison: Placebo vs GB002 (Seralutinib); Test type: Superiority; p = 0.5972, Mixed Models Analysis; Mean Difference (Net) = 6.5, 95% CI 2-sided [-17.9 to 30.9] — GB002 vs. Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Week 28
Arm/Group | Placebo | GB002 (Seralutinib)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 6/42 | 10/44
Other Adverse Events (participants affected / at risk) | 28/42 | 31/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | GB002 (Seralutinib) (N=44)
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 3 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Device malfunction (Product Issues) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | GB002 (Seralutinib) (N=44)
COVID-19 (Infections and infestations) | 7 | 6
Nasopharyngitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Nightmare (Psychiatric disorders) | 1 | 4
Headache (Nervous system disorders) | 8 | 6
Dizziness (Nervous system disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 6 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Fatigue (General disorders) | 3 | 5
Chest discomfort (General disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04456998/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04456998/SAP_001.pdf